CLINICAL TRIAL: NCT05373992
Title: Effect of Exercise and Restrictions to Screen-time on Sport-related Concussion Recovery Time Among Adolescents
Brief Title: Concussion Screen Use Recovery Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Health (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, John Abt, PhD, Andrews Institute Research, Children's Health
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU-2022-0150; ABC (Other: Children's Health Foundation)
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2023-09

CONDITIONS: Sport-related Concussion
Keywords: Concussion; Sports related head injury
MeSH Terms: conditions — Brain Concussion | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Screen Time Restricted (Experimental): Participants will be asked to limit all screen-based activities (television, smartphone, tablet, computer) for the first 72-hours following the initial clinic visit. After the first 72-hours following the initial clinic visit, participants will follow the standard of care as prescribed by their provider. No other specific recommendations will be made to participants regarding exercise, sleep, sedentary time, or physical activity.
  Interventions: Behavioral: Screen Time Restriction (ST-Restricted)
- Aerobic Exercise (Experimental): Participants will be asked to engage in 30-minutes of aerobic exercise (AE) daily for the first 72-hours following the initial clinic visit in the form of a stationary exercise bike, treadmill, or outdoors. The exercise intensity will be prescribed not to exceed 60% of the age-based maximum heart rate. After the first 72-hours following the initial clinic visit, participants will follow the standard of care as prescribed by their provider. No other specific recommendations will be made to participants regarding exercise, sleep, sedentary time, or physical activity.
  Interventions: Behavioral: Aerobic Exercise (AE)
- Screen Time Restricted & Aerobic Exercise (Experimental): Participants will be asked to limit all screen-based activities (television, smartphone, tablet, computer) as well as engage in 30-minutes of AE in the form of a stationary exercise bike, treadmill, or outdoors, for the first 72-hours following the initial clinic visit. The exercise intensity will be prescribed not to exceed 60% of the age-based maximum heart rate. After the first 72-hours following the initial clinic visit, participants will follow the standard of care as prescribed by their provider. No other specific recommendations will be made to participants regarding exercise, sleep, sedentary time, or physical activity.
  Interventions: Behavioral: Screen-time restricted plus aerobic exercise (STR+AE)
- Stretching (Active Comparator): Participants will be asked to follow a daily stretching program for the first 72-hours following the initial clinic visit. After the first 72-hours following the initial clinic visit, participants will follow the standard of care as prescribed by their provider. No other specific recommendations will be made to participants regarding exercise, sleep, sedentary time, or physical activity.
  Interventions: Behavioral: Stretching Only

INTERVENTIONS:
Behavioral: Screen Time Restriction (ST-Restricted) — Participants will be asked to limit all screen-based activities (television, smartphone, tablet, computer) for the first 72-hours following the initial clinic visit. Following the first 72-hours of restricted screen-time, participants will follow the standard of care until the second clinic visit at 7-days post the first clinic visit. No other specific recommendations will be made to participants regarding exercise, sleep, sedentary time, or physical activity.
  Arms: Screen Time Restricted
Behavioral: Aerobic Exercise (AE) — Engage in 30-minutes of aerobic exercise daily for the first 72-hours following the initial clinic visit in the form of a stationary exercise bike, treadmill, or outdoors. The exercise intensity will be prescribed not to exceed 60% of the age-based maximum heart rate (HR). Following the first 72-hours of prescribed AE, participants will follow the standard of care until the second clinic visit at 7-days post the first clinic visit. No other specific recommendations will be made to participants regarding exercise, sleep, sedentary time, or physical activity.
  Arms: Aerobic Exercise
Behavioral: Screen-time restricted plus aerobic exercise (STR+AE) — Participants will be asked to limit all screen-based activities (television, smartphone, tablet, computer) while concurrently engaging in daily aerobic exercise in the form of a stationary exercise bike, treadmill, or outdoors, for the first 72-hours following the initial clinic visit. The exercise intensity will be prescribed not to exceed 60% of the age-based maximum heart rate (HR). Following the first 72-hours of prescribed STR+AE, participants will follow the standard of care until the second clinic visit at 7-days post the first clinic visit. No other specific recommendations will be made to participants regarding exercise, sleep, sedentary time, or physical activity.
  Arms: Screen Time Restricted & Aerobic Exercise
Behavioral: Stretching Only — Participants will be instructed to follow a prescribed stretching program for the first 72-hours following the initial clinic visit. Following the first 72-hours of prescribed stretching, participants will follow the standard of care until the second clinic visit at 7-days post the first clinic visit. No other specific recommendations will be made to participants regarding exercise, sleep, sedentary time, or physical activity.
  Arms: Stretching

SUMMARY:
A two-year parallel randomized clinical trial study to examine the effect of screen time (ST) restriction, exercise alone, and combined ST-restricted-exercise when compared to stretching only (control group) on sports related concussion recovery time among adolescents aged 12 to 17 years. Study hypothesis 1 - There will be significant differences between the treatment and the control arms' mean recovery time (days). Study hypothesis 2 - The ST-restricted & exercise treatment arm will have a significantly shorter mean recovery time (days) compared with the other treatment arms and control arm.

DETAILED DESCRIPTION:
The investigators will randomize a sports related concussion (SRC) treatment protocol (n=313) of Children's Health Andrews Institute for Orthopaedics and Sports Medicine (Andrews) pediatric SRC patients (aged 12-17 years) to one of four treatment groups:1. Screen Time (ST) restricted group, 2.Exercise group, 3.ST restricted & exercise group, and Control [stretching only]) group. The treatments will occur for the first 72-hours following the first clinic appointment. The investigators will monitor treatment adherence and 24-hour movement behaviors over a 72-hour period using the ActiGraph GT9X Link and heart rate monitor; a state-of-the-art research grade wearable device that our research team has expertise in administering and analyzing in field-based studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects
* Age 12-17 years of age presenting to the Children's Health Andrews Institute for Orthopaedics and Sports Medicine (Andrews) concussion clinic in Plano, Texas, to be treated for a diagnosed SRC
* Patients who suffered a sport-related concussion within 72-hours of first clinic visit

Exclusion Criteria:

* Patients who suffered a sport-related concussion outside of 72-hours of first clinic visit
* Is not diagnosed with a SRC
* Is already taking part in another study that measures their physical activity, sleep, screen-time, or is related to concussion
* Has a current diagnosis of and treatment with medication for attention deficit/hyperactivity disorder, learning disorder, depression, anxiety, or a history of more than 3 prior concussions (because these factors are associated with delayed recovery
* Has a co-existing musculoskeletal injury that may impact their ability to be physically active during recovery
* Has an increased cardiac event risk according to the American College of Sports Medicine criteria
* Has a symptom severity score of less than 5 points on the post-concussion symptom scale during the initial clinical examination
* Has an ability to exercise to exhaustion without symptom provocation during the initial clinical examination
* Has limited English language proficiency

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Recovery Time | Day-1 of the participant's self-reported asymptomatic response to unrestricted physical and cognitive activities
  Primary outcome is recovery time (days) as measured as the number of days between the date of injury and day-1 of the participant's self-reported asymptomatic response to unrestricted physical and cognitive activities, which must occur for at least three consecutive days.

SECONDARY OUTCOMES:
Protracted recovery | Greater than 30-days
  Secondary outcome is protracted recovery. A positive classification for protracted recovery is defined as a recovery time, as specified previously, greater than 30-days.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Health - Andrews Institute, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No